CLINICAL TRIAL: NCT01037803
Title: Visualisation of Changes in the Sublingual Microcirculation During Major Surgery Using Sidestream Darkfield Imaging (SDF).
Brief Title: Perioperative Observation of the Sublingual Microcirculation With SDF
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Peter Bentzer, MD, Region Skane
Other Study IDs: USILAN-1
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Surgery
Keywords: perioperative sublingual microcirculation SDF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Does sublingual SDF-imaging results correlate with other haemodynamic parameters measured perioperatively and with postoperative morbidity/complications.

ELIGIBILITY:
Inclusion:

* major surgery > 3h requiring arterial cannulation and central venous access

Exclusion Criteria:

* denied patient consent

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing major surgery at one university hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-10; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bentzer, MD, PhD, Principal Investigator — Dep for Anesthesia and Intensive Care, Lund University Hospital
Locations (1):
- University of Lund and Lund University Hospital, Lund, Skåne County, Sweden